CLINICAL TRIAL: NCT04772781
Title: National, Multicentre, Randomized, Double-blind, Double-dummy Phase II Clinical Trial to Evaluate the Efficacy and Safety of S (+) - Ibuprofen for Pain Control in Individuals With At Least Moderate Mechanical Acute Low Back Pain
Brief Title: Efficacy and Safety of S (+) - Ibuprofen in the Treatment of Mechanical Low Back Pain
Acronym: APS002/2020
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Apsen Farmaceutica S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APS002/2020
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-02

CONDITIONS: Low Back Pain, Mechanical; Low Back Pain; Acute Low Back Pain
Keywords: Pain control; Low back pain; Pain relief; Ibuprofen; Inflammation; Anti-inflammatory
MeSH Terms: conditions — Low Back Pain; Agnosia; Inflammation | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S (+) - Ibuprofen (Experimental)
  Interventions: Drug: S (+) - Ibuprofen
- Ibuflex® - ibuprofen (Active Comparator)
  Interventions: Drug: Ibuflex®

INTERVENTIONS:
Drug: S (+) - Ibuprofen — S (+) - Ibuprofen + placebo of Ibuflex®
  Arms: S (+) - Ibuprofen
Drug: Ibuflex® — Ibuflex® + placebo of S (+) - Ibuprofen
  Arms: Ibuflex® - ibuprofen

SUMMARY:
The purpose of this study is to evaluate the efficacy of S (+) - ibuprofen compared to an active treatment for pain control in individuals with at least moderate acute mechanical low back pain.

ELIGIBILITY:
Main Inclusion Criteria:

* Ability to confirm voluntary participation and agree to all trial purposes by signing and dating the informed consent forms;
* Patient with acute low back pain who responds to the pain period less than or equal to 3 days;

Main Exclusion Criteria:

* Known hypersensitivity to the formula components used during the clinical trial;
* Previous history of alcohol or drugs abuse diagnosed by DSM-V;
* Current or previous history (less than 12 months) of smoking;
* Have clinically relevant abnormal laboratory results according to medical evaluation;
* Women who are pregnant, lactating, or positive for β - hCG urine test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
At least 50% of maximum pain relief score in Maximum Total Pain Relief (TOTPARmax) | Change from Baseline to 6 hours
  TOTPAR was calculated using data from a 5-point categorical pain relief scale (none = 0, slight = 1, moderate = 2, good = 3, or complete pain relief = 4)

SECONDARY OUTCOMES:
Adverse events rates between groups | During treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Apsen Farmacêutica S.A., São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No